CLINICAL TRIAL: NCT03063762
Title: An Open-Label, Multi-Center, Randomized, Dose-Escalation, Phase 1b Study to Evaluate Safety, Pharmacokinetics and Therapeutic Activity of RO6874281 in Combination With Atezolizumab ± Bevacizumab in Patients With Unresectable Advanced and/or Metastatic Renal Cell Carcinoma
Brief Title: Study to Evaluate Safety, Pharmacokinetics and Therapeutic Activity of RO6874281 as a Combination Therapy in Participants With Unresectable Advanced and/or Metastatic Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP39365; 2016-003528-22 (EudraCT Number)
Record Dates: First submitted 2017-02-22; First posted 2017-02-24 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; RO6874281; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Escalation Part (Arm A): Atezolizumab, RO6874281 (Experimental): Participants will receive RO6874281 in combination with atezolizumab once a week for 4 weeks followed by once every 2 weeks afterwards until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has complete response (CR), treatment may be discontinued and reintroduced if progressive disease (PD), for a maximum duration of 24 months.
  Interventions: Drug: Atezolizumab; Drug: RO6874281
- Escalation Part (Arm B): Atezolizumab, Bevacizumab, RO6874281 (Experimental): Participants will receive RO6874281 in combination with atezolizumab and bevacizumab until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has CR, treatment may be discontinued and reintroduced if PD, for a maximum duration of 24 months.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: RO6874281
- Extension Part (Arm A): Atezolizumab, RO6874281 (Experimental): Based on the maximum tolerated dose or recommended dose as determined in the dose-escalation part, participants will receive RO6874281 in combination with atezolizumab once a week for 4 weeks followed by once every 2 weeks afterwards until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has CR, treatment may be discontinued and reintroduced if PD, for a maximum duration of 24 months.
  Note: no new participants are being enrolled in the arm at this time.
  Interventions: Drug: Atezolizumab; Drug: RO6874281
- Extension Part (Arm B): Atezolizumab, Bevacizumab, RO6874281 (Experimental): Based on the maximum tolerated dose or recommended dose as determined in the dose-escalation part, participants will receive RO6874281 in combination with atezolizumab and bevacizumab once a week for 4 weeks followed by once every 2 weeks afterwards until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has CR, treatment may be discontinued and reintroduced if PD, for a maximum duration of 24 months.
  Note: no new participants are being enrolled in the arm at this time.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: RO6874281
- Extension Part (Arm C): Atezolizumab, RO6874281 (Experimental): Based on the maximum tolerated dose or recommended dose as determined in the dose-escalation part, participants will receive RO6874281 in combination with atezolizumab once every 3 weeks until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has CR, treatment may be discontinued and reintroduced if PD, for a maximum duration of 24 months.
  Note: no new participants are being enrolled in the arm at this time.
  Interventions: Drug: Atezolizumab; Drug: RO6874281
- Extension Part (Arm D): Atezolizumab, Bevacizumab, RO6874281 (Experimental): Based on the maximum tolerated dose or recommended dose as determined in the dose-escalation part, participants will receive RO6874281 in combination with atezolizumab and bevacizumab once every 3 weeks until disease progression, unacceptable toxicities, or withdrawal of consent, or as long as the participant experiences clinical benefit, or if the participant has CR, treatment may be discontinued and reintroduced if PD, for a maximum duration of 24 months.
  Note: Arm D is closed for future enrollment
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: RO6874281

INTERVENTIONS:
Drug: Atezolizumab — Arms A and B Atezolizumab will be administered at a dose of 840 milligrams (mg) prior to RO6874281 administration as an intravenous (IV) infusion on Days 1, 15, 29, and once in 2 weeks from Day 29 onwards. Doses in the extension part will be based on the maximum tolerated dose determined in the escalation part.
  Arms C and D Atezolizumab will be administered at a dose of 1200mg as it is a Q3W schedule
  Other Names: Tecentriq®
Drug: Bevacizumab — Arms A and B Bevacizumab will be administered at a dose of 10 milligrams per kilogram (mg/kg) after the atezolizumab administration, and prior to RO6874281 administration as an IV infusion on Days 15, 29, and once in 2 weeks from Day 29 onwards.
  In Arm D, Bevacizumab will be administered at a dose of 15mg/kg on Day 8 of Cycle 2 and on Day 8 of each consecutive cycle.
  Other Names: Avastin®
  Arms: Escalation Part (Arm B): Atezolizumab, Bevacizumab, RO6874281; Extension Part (Arm B): Atezolizumab, Bevacizumab, RO6874281; Extension Part (Arm D): Atezolizumab, Bevacizumab, RO6874281
Drug: RO6874281 — Arms A and B RO6874281 will be administered as an IV infusion on Days 1, 8, 15, 22, and 29, and once in 2 weeks from Day 29 onwards. Starting dose of RO6874281 will be 5 mg, and will be increased subsequently. Doses in the extension part will be based on the maximum tolerated dose determined in the escalation part.
  In Arms C and D, RO will be administered on Q3W schedule at the dose defined in the dose escalation part
  Other Names: simlukafusp alfa

SUMMARY:
This is an open-label, multi-center, randomized, Phase 1b, adaptive, clinical study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary therapeutic activity of RO6874281 in combination with atezolizumab with/without bevacizumab in participants with unresectable advanced and/or metastatic RCC. The study will consist of a dose-escalation part and an extension part.

ELIGIBILITY:
Inclusion criteria:

* Unresectable advanced and/or metastatic RCC with component of clear cell histology and/or component of sarcomatoid histology that has not been previously treated with any systemic therapy, including treatment in the adjuvant setting
* During dose escalation only, an additional population with unresectable advanced and/or metastatic 2nd line RCC patients is allowed
* At least one tumor lesion with location accessible to biopsy per clinical judgment of the treating physician
* Consent to provide an archival tumor tissue sample (if available) and to undergo baseline and on treatment tumor biopsies for pharmacodynamic biomarker analysis
* Measurable disease, as defined by RECIST v1.1. At least one lesion accessible for biopsy
* Participants with unilateral pleural effusion are eligible if they fulfill both of the following: (a) New York Heart Association (NYHA) Class 1; (b) Global initiative for obstructive lung disease (GOLD) test level 1 (forced expiratory volume in 1 second [FEV1]/ forced vital capacity [FVC] less than [<] 0.7 and FEV1 greater than or equal to [>=] 80 percent [%] predicted after inhaled bronchodilator)

Adequate hematological function: neutrophil count of ≥1.5 ≥109 cells/L, platelet count of ≥100,000/≥L, Hb ≥9 g/dL (5.6 mmol/L), lymphocytes ≥0.8 ≥109 cells/L.

Exclusion Criteria:

* Symptomatic or untreated central nervous system (CNS) metastases
* Participants with asymptomatic CNS metastases with previous or concomitant brain deficiencies, as defined in the protocol
* Participants with confirmed bilateral pleural effusion
* Episode of significant cardiovascular/cerebrovascular acute disease within 6 months prior to Cycle 1 Day 1
* Active or uncontrolled infections
* Human immunodeficiency virus (HIV) or active Hepatitis A, B, C, D and E virus (HAV, HBV, HCV, HDV and HEV) infection.
* Major surgery or significant traumatic injury <28 days prior to Cycle 1 Day 1 (excluding fine needle biopsies) or anticipation of the need for major surgery during study treatment
* Serious, non-healing wound; active ulcer; or untreated bone fracture
* Proteinuria as demonstrated by a urine protein to creatinine ratio (UPCR) of >=1.0 at screening
* History of, active or suspicion of autoimmune disease
* Concurrent use of high dose of systemic steroids. The use of inhaled, topical and ophthalmic steroids is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Arm A: It ends one week after the second administration of RO6874281 + atezolizumab Arm B: one week after the first administration of RO6874281 + atezolizumab + bevacizumab
  The first patient in each cohort and regimen will be observed for safety for one week after the administration of RO6874281and atezolizumab +-bevacizumab, prior to enrollment of additional patients in a cohort.
  The DLT will be counted for each dose separately and each patient will contribute one single representative data point.
Maximum Tolerated Dose (MTD) of RO6874281 | Arm A: It ends one week after the second administration of RO6874281 + atezolizumab Arm B: one week after the first administration of RO6874281 + atezolizumab + bevacizumab
  The MTD is defined as the highest dose with less than 33% probability of dose limiting toxicity (DLT).
Recommended Dose of RO6874281 | Arm A: It ends one week after the second administration of RO6874281 + atezolizumab Arm B: one week after the first administration of RO6874281 + atezolizumab + bevacizumab
  The recommended dose is defined as the lowest safe dose with the best likelihood for clinical benefit.
Percentage of Participants with Objective Response of Complete Response (CR) or Partial Response (PR) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Screening until disease progression or study treatment discontinuation (assessed at every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 24 months)
  Objective response rate (ORR) defined as the number of patients who achieved an objective response (partial response (PR) plus complete response (CR)) confirmed 28 or more days later, as determined by the Investigator using RECIST v1.1 and modified RECIST criteria at any time during the study divided by the number of response-evaluable patients.

SECONDARY OUTCOMES:
Serum RO6874281 Concentration | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 1 hour (hr) post start of infusion, end of infusion (EOI), 2, 6 hr post EOI on Cycle 1 Day 1; Cycle 1 Days 2, 3; Pre-infusion, 1 hr post start of infusion, EOI, 2, 6 hr post EOI on Cycle 1 Day 8; Cycle 1 Days 9, 10; Pre-infusion, EOI on Cycle 2 Day 1; Pre-infusion on Cycle 3 Day 1; Cycle 3 Day 2; Pre-infusion on Cycle 4 Day 1; Pre-infusion on Cycle 5 Day 1; Cycle 5 Day 2; Pre-infusion on Day 1; Day 2 in Cycle 9 and then every 4 cycles for the first year followed by every 6 cycles; treatment discontinuation; 28 days after last dose; 3 months after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 1, 2; -4 hr for other timepoints) (infusion length = 2 hr) (1 cycle = 15 days)
Area Under the Serum Concentration-Time Curve (AUC) for RO6874281 | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 1 hr post start of infusion, EOI, 2, 6 hr post EOI on Cycle 1 Day 1; Cycle 1 Days 2, 3; Pre-infusion, 1 hr post start of infusion, EOI, 2, 6 hr post EOI on Cycle 1 Day 8; Cycle 1 Days 9, 10; Pre-infusion, EOI on Cycle 2 Day 1; Pre-infusion on Cycle 3 Day 1; Cycle 3 Day 2; Pre-infusion on Cycle 4 Day 1; Pre-infusion on Cycle 5 Day 1; Cycle 5 Day 2; Pre-infusion on Day 1; Day 2 in Cycle 9 and then every 4 cycles for the first year followed by every 6 cycles; treatment discontinuation; 28 days after last dose; 3 months after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 1, 2; -4 hr for other timepoints) (infusion length = 2 hr) (1 cycle = 15 days)
Maximum Observed Serum Concentration (Cmax) of RO6874281 | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 1 hr post start of infusion, EOI, 2, 6 hr post EOI on Cycle 1 Day 1; Cycle 1 Days 2, 3; Pre-infusion, 1 hr post start of infusion, EOI, 2, 6 hr post EOI on Cycle 1 Day 8; Cycle 1 Days 9, 10; Pre-infusion, EOI on Cycle 2 Day 1; Pre-infusion on Cycle 3 Day 1; Cycle 3 Day 2; Pre-infusion on Cycle 4 Day 1; Pre-infusion on Cycle 5 Day 1; Cycle 5 Day 2; Pre-infusion on Day 1; Day 2 in Cycle 9 and then every 4 cycles for the first year followed by every 6 cycles; treatment discontinuation; 28 days after last dose; 3 months after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 1, 2; -4 hr for other timepoints) (infusion length = 2 hr) (1 cycle = 15 days)
Serum Atezolizumab Concentration | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 1 Day 1; Pre-infusion on Cycle 1 Day 8; Pre-infusion on Day 1 Cycles 2, 3, 4, 5, and 9 onwards; treatment discontinuation; 28, 120 days after last dose (up to 60 months) (Pre-infusion = -4 hr) (infusion length = 1 hr) (1 cycle = 15 days)
AUC of Atezolizumab | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 1 Day 1; Pre-infusion on Cycle 1 Day 8; Pre-infusion on Day 1 Cycles 2, 3, 4, 5, and 9 onwards; treatment discontinuation; 28, 120 days after last dose (up to 60 months) (Pre-infusion = -4 hr) (infusion length = 1 hr) (1 cycle = 15 days)
Cmax of Atezolizumab | Pre-infusion on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 1 Day 1; Pre-infusion on Cycle 1 Day 8; Pre-infusion on Day 1 Cycles 2, 3, 4, 5, and 9 onwards; treatment discontinuation; 28, 120 days after last dose (up to 60 months) (Pre-infusion = -4 hr) (infusion length = 1 hr) (1 cycle = 15 days)
Serum Bevacizumab Concentration | Pre-infusion on Cycle 2 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 2 Day 1; Pre-infusion on Cycle 2 Day 8; Pre-infusion on Day 1 Cycles 3, 4, 5, and 9 onwards; treatment discontinuation; 28 days after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 2, 3; -4 hr for other timepoints) (infusion length = 1.5 hr) (1 cycle = 15 days)
AUC of Bevacizumab | Pre-infusion on Cycle 2 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 2 Day 1; Pre-infusion on Cycle 2 Day 8; Pre-infusion on Day 1 Cycles 3, 4, 5, and 9 onwards; treatment discontinuation; 28 days after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 2, 3; -4 hr for other timepoints) (infusion length = 1.5 hr) (1 cycle = 15 days)
Cmax of Bevacizumab | Pre-infusion on Cycle 2 Day 1 up to 60 months (detailed timeframe is provided in outcome measure description)
  Pre-infusion, 0.5 hr post EOI on Cycle 2 Day 1; Pre-infusion on Cycle 2 Day 8; Pre-infusion on Day 1 Cycles 3, 4, 5, and 9 onwards; treatment discontinuation; 28 days after last dose (up to 60 months) (Pre-infusion = 0 hr for Day 1 Cycles 2, 3; -4 hr for other timepoints) (infusion length = 1.5 hr) (1 cycle = 15 days)
Percentage of Participants with Anti-Drug Antibodies (ADA) to RO6874281 | Baseline until 3 months post last dose of study treatment (detailed timeframe is provided in outcome measure description)
  Baseline until 3 months post last dose of study treatment (assessed at pre-infusion on Days 1, 8 of Cycle 1; Pre-infusion on Day 1 of Cycles 2, 3, 4, 5, 9 and then every 4 cycles for the first year followed by every 6 cycles; treatment discontinuation; 28 days after last dose; 3 months after last dose [up to 60 months] [Pre-infusion = 0 hr for Day 1 Cycles 1, 2; -4 hr for other timepoints] [infusion length = 2 hr] [1 cycle = 15 days])
Absolute Lymphocytes Count in Peripheral Blood | Screening until 120 days post last dose of study treatment (up to 60 months)
  At baseline; Day 1, 2 3, 8 of Cycle 4. Day 1, 2 of Cycle 5 and Cycle 6. Day 1 of Cycle 7, Cycle 8 and Subsequent Cycles; At treatment discontinuation; 28 days after last dose; 3 months after last dose
Density of Lymphocytes in Tumor Samples | Archival biopsy: Baseline; Fresh biopsies: Baseline, Day 8 of Cycle 4; Optional biopsies: Any time during the study conduct (1 cycle = 15 days) (up to 60 months)
Percentage of Participants with Programmed Death-Ligand 1 (PD-L1) Status in Tumor Samples | Archival biopsy: Baseline; Fresh biopsies: Baseline, Day 8 of Cycle 4; Optional biopsies: Any time during the study conduct (1 cycle = 15 days) (up to 60 months)
Percentage of Participants with CR as Determined by the Investigator Using RECIST v1.1 | Screening until disease progression or study treatment discontinuation (assessed at every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 24 months)
Percentage of Participants with Disease Control as Determined by the Investigator Using RECIST v1.1 | Screening until disease progression or study treatment discontinuation (assessed at every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 24 months)
Duration of Response (DOR) as Determined by the Investigator Using RECIST v1.1 | Screening until disease progression or study treatment discontinuation (assessed at every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 24 months)
Progression-Free Survival (PFS) as Determined by the Investigator Using RECIST v1.1 | From randomization until disease progression or study treatment discontinuation (assessed at every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 24 months)
Overall Survival (OS) | From randomization until death (up to 60 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (3):
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Northwestern Center for Clinical Research; Cancer Center, Chicago, Illinois
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Herlev Hospital; Afdeling for Kræftbehandling, Herlev, Denmark
- France (2):
  - Centre Léon Bérard - Centre régional de lutte contre le cancer Rhône-Alpes, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
- Germany (2):
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
  - Uniklinikum, Comprehensive Cancer Center Mainfranken; Interdisziplinäres Studienzentrum mit ECTU, Würzburg
- Italy (2):
  - Universita di Modena e Reggio Emilia;Dipartimento di Oncologia ed Ematologia, Modena, Emilia-Romagna
  - Fondazione IRCCS Policlinico San Matteo, Oncologia, Pavia, Lombardy
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- United Kingdom (3):
  - Barts & London School of Med; Medical Oncology, London
  - The Christie, Manchester
  - Southampton General Hospital; Medical Oncology, Southampton